CLINICAL TRIAL: NCT02058810
Title: Does the Use of Optiflow High Flow Oxygen on Patients With Acute Cardial Decompensation (NYHA Classification Stage III-IV) Allow for Quicker Improvement of the Organ Dysfunction Than Conventional Standard-Oxygen-Insufflation-Therapy?
Brief Title: Nasal High Flow at Acute Hart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients, PI left
Sponsor: University Hospital Regensburg (Other)
Collaborators: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Maximilian Malfertheiner, Dr. med, University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300513
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Decompensated Heartfailure; Cardio-renal Syndrom
Keywords: nasal high flow oxygen; cardio-renal syndrom; heartfailure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional nasal Oxygen (Other): Conventional nasal Oxygen as needed
  Interventions: Device: Conventional nasal oxygen
- Nasal high flow (Other): Nasal high flow therapy with FiO2 40% and flow of 40l/min for at least 48h
  Interventions: Device: Nasal high flow

INTERVENTIONS:
Device: Nasal high flow
  Other Names: Optiflow; Fisher & Paykel Healthcare; RT202
  Arms: Nasal high flow
Device: Conventional nasal oxygen
  Other Names: nasal oxygen
  Arms: Conventional nasal Oxygen

SUMMARY:
The pilot study aims to compare the results of using a new respirator (OPTIFLOW TM-High-Flow-Machine) with those from Standard-Oxygen-Therapy during the stabilization of patients who have been hospitalized due to acute heart failure. We expect a faster and more effective stabilization after acute cardial decompensation among the patients with the High-Flow-machine.

The study should show whether the use of High-Flow-Therapy leads to a relevant improvement in terms of objective clinical parameters of heart failure like those for cardial-renal syndrome, changes in the nt-pro-BNP, weight loss, changes in the diameter of the inferior vena cava, in terms of the degree of shortness of breath and decompensation, and whether subjective clinical symptoms like dyspnea and quality of life differ between the two groups of patients.

The investigators see the primary outcome of the study as the improvement of the cardial-renal syndrome as a sign of the more effective stabilisation compared to the standard therapy. Furthermore, the investigators expect a quicker decrease in serum creatinine and an improvement in the creatinine clearance through therapy with the High-Flow-Machine. In terms of secondary outcomes of the study, the investigators are interested in also comparing e.g., the duration of hospital stays, 90-day mortality, and rehospitalisation within three months. Here, the investigators expect a quicker improvement in the subjective shortness of breath of the patients who are treated using the Hifh-Flow-Machine. Moreover, we believe that along with the individual subjective improvements (quality of life survey), the patients will experience a quicker release from the hospital and in this way, lead to a healthcare economic improvement among patients with repeated hospitalizations who usually have chronic problems.

It is also of great interest to us, whether the biomarker BNP is an appropriate parameter for determining the faster stabilization of the patient and whether the degree of improvement of subjective dyspnea is correlated with the time needed until the patient has been stabilised.

DETAILED DESCRIPTION:
Primary endpoint:

Improvement of the cardiorenal syndrome type1 measured by the improvement of creatine clearance and the Serum-Creatinin of patients undergoing High-Flow treatment.

Secondary endpoints:

Worsening of cardiac insufficiency (application of catecholamines, need of NIV, intubation, death) Duration of hospital stay (in days) 90-day mortality Readmittance to hospital within 3 months Intrathoracic bloodvolume at hospital discharge Change of dyspnea at 3h, 6h, 24h > VAS-0-100 (visual analog scale) Change in the diameter of the IVC (inferior vena cava) as a non-invasive parameter for assessing the degree of decompensation Change in the BNP (hospital admission vs. discharge, after 3 months) Weight loss in hospital Amount of diuretics

ELIGIBILITY:
Inclusion Criteria:

* patients with acute heartfailure NYHA III und IV

Exclusion Criteria:

* Patients wit respiratory insufficency and indication for mechanical ventilation
* Asthma bronchiale
* severe COPD
* cardiogenic shock (RR persisting< 90mmHg systolic or catecholamine application)
* renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cardiorenal syndrome type 1 | 3 Months
  The acute deterioration of the cardial situation often leads to a consecutive deterioration of renal function. The damage to renal function caused by acute cardial genesis is defined as cardiorenal syndrome type 1 [2]. In such cases, the venous congestion with heightened central venous pressure leads to disruption of renalfunction and possibly even to acute kidney failure [3, 4]. This is defined as cardiorenal syndrom with an increase in serumcreatine of >0,3 mg/dl and is associated with higher mortality and longer hospital stays [5].

SECONDARY OUTCOMES:
Change of dyspnea | 3h, 6h, 24h
  Change of dyspnea at 3h, 6h, 24h > VAS-0-100 (visual analog scale)

OTHER OUTCOMES:
90-day mortality | 90 days
  Mortality after 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- UHMagdeburg, Magdeburg, Saxony-Anhalt, Germany